CLINICAL TRIAL: NCT06965504
Title: Initiation and Titration of Guideline Directed Medical Therapy in Heart Failure Cardiogenic Shock With Impella 5.5 for Cardiac Recovery: INTeGRATE
Brief Title: INitiation and Titration of Guideline Directed Medical TheRApy in HearT Failure Cardiogenic Shock With ImpElla 5.5 for Cardiac Recovery
Acronym: INTeGRATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTeGRATE
Record Dates: First submitted 2025-04-21; First posted 2025-05-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Cardiogenic Shock; Reduced Ejection Fraction Heart Failure
Keywords: Impella 5.5; Heart Failure Cardiogenic Shock; Reduced Ejection Fraction Heart Failure; Mechanical Circulatory Support; Cardiovascular Disease; Heart Disease; Guideline Directed Medical Therapy
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic; Heart Failure, Systolic; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study (Other): This is a single arm study.
  Interventions: Device: Impella 5.5 SmartAssist

INTERVENTIONS:
Device: Impella 5.5 SmartAssist — The intervention is Impella 5.5 with SmartAssist® support combined with heart failure guideline directed medical therapy (GDMT).

SUMMARY:
The study will evaluate if Impella 5.5® support in heart failure reduced ejection fraction (HFrEF) patients presenting with decompensated heart failure (HF) and cardiogenic shock will facilitate the initiation and optimization of guideline directed medical therapy (GDMT) during the hospital stay and post-discharge.

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-center, post-market, on-label study. Patients presenting with HFrEF who are not on adequate GDMT and who are presenting with heart failure cardiogenic shock will be evaluated for inclusion. The study objectives are to evaluate the impact of Impella 5.5 support on GDMT up-titration during support, at discharge, and at 90-days post-discharge and to evaluate the feasibility of Impella 5.5 combined with optimal GDMT to improve heart recovery in patients with decompensated heart failure. Outcomes will be measured up to one-year post-hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and < 75 years
2. Subject has signed the Informed Consent
3. LVEF ≤ 40%
4. History of HF <5 years
5. Subject is presenting with decompensated heart failure and meets one of the following cardiogenic shock criteria:

   1. Sustained episode of systolic blood pressure ≤ 90 mmHg for at least 30 minutes or need for vasoactive agents to maintain such blood pressure.
   2. Or serum lactate > 2 mmol/L
   3. Or a cardiac index (CI) < 2.2 L/min/m2 determined to be secondary to cardiac dysfunction, in the absence of hypovolemia
   4. Or required support with an intra-aortic balloon pump (IABP)
6. Subject has inadequate heart failure GDMT based on the most recent outpatient prescription prior to index admission as determined by the treating cardiologist and the Eligibility Committee, defined as:

   1. On 2 or less of the evidence-based GDMT (BB, MRA, SGLT2i, and RASi)
   2. If on β-blocker and RASi, at least one of the two medications is <50% of maximal dose.

Exclusion Criteria:

1. Underlying unmodifiable conditions that limit initiation of GDMT prior to enrollment, including but not limited to:

   1. Drug allergies or hypersensitivities to HF GDMT medications, unless alternative can be identified.

      Drug allergy/hypersensitivity is an immune-mediated reaction to a medication. Adverse reactions must be a result of immune or inflammatory cell stimulations by the mеԁiсаtion:
   2. Known bilateral renal artery stenosis
   3. Type 1 diabetes
   4. 2nd or 3rd degree AV block, unless pacemaker is in place
   5. Angioedema, hereditary or idiopathic
   6. Pregnancy, known or confirmed by a pregnancy test if of child bearing potential.
2. Cardiogenic shock due to myocardial infarction prior to enrollment
3. Mixed shock, septic shock, or shock from non-cardiac origins
4. Severe Cardiogenic Shock, defined as meeting one or more of the below prior to enrollment:

   1. SCAI stage E per Study Definition (Appendix C)
   2. Serum lactate > 8mmol/L
   3. On mechanical circulatory support (not including IABP) or on mechanical ventilation for non-procedural reasons.
   4. Experiencing pulseless electrical activity (PEA) or refractory ventricular tachycardia (VT)/ventricular fibrillation (VF)
   5. Severe acidosis (pH < 7.2 or bicarbonate < 10mEq/L)
5. In cardiac arrest prior to enrollment
6. Revascularization or cardiac surgery within 90-days of the index hospitalization date or decision to undergo revascularization or cardiac surgery made prior to enrollment.
7. Inflammatory and infiltrative cardiomyopathy (CM) including myocarditis, restrictive CM, constrictive pericarditis, or hypertrophic CM including sarcoidosis and amyloidosis.
8. Adult congenital heart disease without appropriate surgical correction
9. Structural or anatomical abnormalities that cannot be modified as determined by the treating cardiologist, including severe primary mitral regurgitation (MR) .
10. Severe RV dysfunction, per Study Definition (Appendix C), requiring mechanical or inotropic support prior to enrollment.
11. Severe dilatation of the LV with LVEDD greater than 8.0cm
12. History of heart transplant or listed for heart transplant prior to enrollment.
13. Planned to be implanted with a permanent VAD within 90-days of the index hospitalization date.
14. Continuous outpatient inotropic support prior to the index hospitalization date.
15. Planned to pursue palliative care or hospice, or life expectancy of less than 2 years due to non-cardiac illness at the time of index hospitalization date.
16. ICD upgrade to BiV, or implantation of CRT within 30-days of the index hospitalization date.
17. Currently on dialysis, or has pre-existing end-stage chronic kidney disease (stage 4 or above), or has hereditary, infectious, or autoimmune nephropathy.
18. Pre-existing liver dysfunction defined as: presence of liver cirrhosis or alcoholic hepatitis, or presence of acute liver failure or acute hepatitis not due to cardiogenic shock.
19. Pre-existing pulmonary disease requiring home oxygen
20. History of stroke or intracranial hemorrhage ≤ 90 days of the index hospitalization date, or a history of cerebrovascular disease with significant (> 80%) uncorrected carotid stenosis, or any permanent neurological deficit with mRS score >2.
21. Any contraindication that precludes placing an Impella 5.5®, including but not limited to:

    1. Aortic valve stenosis/calcification with orifice area ≤0.6cm2 or aortic insufficiency of any grade greater than mild on pre-procedure echocardiography.
    2. Presence of mechanical aortic valve or heart constrictive device.
    3. Thrombus in the left atrium or ventricle.
    4. Infection of the planned procedural access site or suspected systemic active infection.
    5. Severe arterial disease precluding placement of Impella.
    6. Presence of Atrial or Ventricular Septal Defect (including post-infarct VSD)
    7. Left ventricular rupture
    8. Cardiac tamponade I. Combined cardiorespiratory failure
22. Known contraindication to heparin (i.e., heparin induced thrombocytopenia (HIT)) or intolerance to anticoagulant or antiplatelet therapies.
23. Allergies or contraindications to contrast agents unless can be adequately medicated.
24. History of bleeding diathesis or known coagulopathy, any GU or GI bleed within 90-days of the index hospitalization date or will refuse blood transfusions.
25. Subject has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures.
26. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device that has not met its primary endpoint.
27. Subject belongs to a vulnerable population, such as such as prisoners, individuals with impaired decision making, or economically or educationally disadvantaged persons.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
% of Subjects achieving indicated GDMT treatment | Hospital discharge
  Achieving any dose of all four GDMT classes

OTHER OUTCOMES:
% of Subjects achieving optimized GDMT treatment | Through 1-year post-discharge
  Achieving any dose of all four classes and at least 50% of the target dose of β-blocker and RASi
Modified Heart Failure Collaboratory (mHFC) score | Through 1-year post-discharge
  Defined by HFC in 2022. Improvement from baseline
Rate of GDMT-Related Serious Adverse Events | Through 1-year post-discharge
  The composite rate of any of the following GDMT-related serious adverse events:
  1. Recurrence or worsening shock; symptomatic hypotension requiring admission
  2. Bradycardia requiring treatment
  3. Hyperkalemia requiring intervention
  4. Ketoacidosis requiring treatment
  5. Need for new renal replacement therapy (RRT)
% of Subjects free from heart replacement | Through 1-year post-discharge
  Freedom from durable ventricular assist device (VAD) or heart transplant (HTx)
Rate of subjects with HF hospitalization or urgent HF visit | Through 1-year post-discharge
% of Subjects with cardiovascular mortality and all cause mortality | Through 1-year post-discharge
% of Subjects with all-cause death | Through 1-year post-discharge
Left ventricular ejection fraction (LVEF) | Through 1-year post-discharge
  Change from baseline
Left ventricular end-diastolic diameter (LVEDD) | Through 1-year post-discharge
  Change from baseline
N-Terminal pro b-type natriuretic peptide (NT-proBNP) | Through 1-year post-discharge
  Change from baseline
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Through 1-year post-discharge
  Improvement from baseline
Quality of life assessed by EuroQoL 5-Dimensions 5-Levels (EQ-5D-5L) | Through 1-year post-discharge
  Improvement from baseline
6-Minute Walk Test Distance | Through 1-year post-discharge
  Improvement from baseline
New York Heart Association (NYHA) heart failure class | Through 1-year post-discharge
  Improvement from baseline
Society for Cardiovascular Angiography & Interventions (SCAI) shock stage | Time of device removal
  Improvement from baseline
Rate of major device-related adverse events | Hospital discharge
  The composite rate of any of the following device-related serious adverse events:
  1. Major vascular access site complication
  2. Major hemolysis
  3. Bleeding, defined as MCS-ARC Type 3 or higher
  4. Structural complication requiring repair
  5. Stroke
GDMT Optimization Change Score | Through 1-year post-discharge
  Sum of positive therapy changes (+2 for new GDMT initiations, +1 for dose uptitration) and negative therapy changes (-2 for GDMT discontinuation, -1 for dose downtitration) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Adam DeVore, MD, MHS, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Tampa General Hospital, Tampa, Florida
  - Abbott Northwestern, Minneapolis, Minnesota
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Centennial Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No